CLINICAL TRIAL: NCT05312099
Title: The Effect of Menopause on Sexual Life and Depression: a Case-control Study.
Acronym: menopause
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Research assistant, Hitit University
Other Study IDs: 2018-20
Record Dates: First submitted 2021-12-03; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Menopause; Depression; Sexual Dysfunction
MeSH Terms: conditions — Depression; Sexual Dysfunction, Physiological | interventions — Case-Control Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Women who have entered early menopause (before the age of 40), have chronic systemic diseases (diabetes, heart disease, hypertension, thyroid, rheumatic disease, psychiatric disease history), and use psychiatric drugs were not included in the study.
  Interventions: Other: Case control
- Control group: Women under the age of 45, over the age of 55 with chronic systemic diseases (diabetes, heart disease, hypertension, thyroid, rheumatic disease, psychiatric disease history) and using psychiatric drugs were not included in the study.
  Interventions: Other: Case control

INTERVENTIONS:
Other: Case control — Case control study

SUMMARY:
work completed but not yet published

DETAILED DESCRIPTION:
work completed but not yet published

ELIGIBILITY:
Inclusion Criteria:

* Case group: Women between the ages of 45-65, who are in the postmenopausal period, who are literate, who do not have communication difficulties / mental disabilities, and who volunteer to participate in the study were included.

Control Group: Women between the ages of 45-55, who were not menopausal, who were literate, who had no communication difficulties / mental disabilities and who volunteered to participate in the study were included.

Exclusion Criteria:

* For case group: Women with premature menopause (before the age of 40), chronic systemic disease (diabetes, heart disease, hypertension, thyroid, rheumatic disease, psychiatric disease history) and using psychiatric drugs were not included in the study.

For control group: Women under the age of 45, over the age of 55 with chronic systemic diseases (diabetes, heart disease, hypertension, thyroid, rheumatic disease, psychiatric disease history) and using psychiatric drugs were not included in the study.

Ages: 45 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Çorum Hitit University Erol Olçok Training and Research Hospital Obstetrics and Gynecology Policlinic was composed of 200 married women between the ages of 45-65, 113 of them in the postmenopausal period and 87 of them did not go through menopause.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
The effect of menopause on sexual life and depression: a case-control study. | 14.01.2019-16.02.2021
  Data completed in April 2019

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Yıldırım, Principal Investigator — Fatma
Locations (1):
- Hitit university, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No